CLINICAL TRIAL: NCT02664857
Title: Effect of Vitamin D Supplementation on Postoperative Pain and Sedation-agitation
Brief Title: Vitamin D Supplementations and Postoperative Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, ebru biricik, Medical Doctor, Cukurova University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Vitamin D
Record Dates: First submitted 2016-01-20; First posted 2016-01-27 (Estimated); Last update posted 2021-04-21 (Actual); Status verified 2021-01

CONDITIONS: Postoperative Pain
Keywords: Vitamin D; Postoperative Pain; Mental Motor Retardation
MeSH Terms: conditions — Pain, Postoperative | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- vitamin D (Active Comparator): After per orally vitamin D supplementation during 12 weeks, serum Vitamin D level will evaluate with laboratory testing. 600 IU vitamin D will apply to 30 subject during 12 weeks. At first day end end of the 12 weeks serum vitamin D level will analyse with laboratory testing.End of the 12 weeks, the children will be perform dental treatment under general anaesthesia. Postoperative pain, anxiety and sedation will evaluate.
  Interventions: Drug: Vitamin D
- Placebo (Sham Comparator): Grup P will not take vitamin D during 12 weeks. This group just only will follow by researchers.At first day end end of the 12 weeks serum vitamin D level will analyse with laboratory testing.End of the 12 weeks, the children will be perform dental treatment under general anaesthesia. Postoperative pain, anxiety and sedation will evaluate.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D — Group D will take 600 IU vitamin D per orally during 12 weeks. At first day and end of the 12 weeks serum vitamin D level will analyse with laboratory testing
  Other Names: vitamin D supplementation
  Arms: vitamin D
Drug: Placebo — Group P will not take orally during 12 weeks. This group will only observe by researchers.
  Other Names: Observed group
  Arms: Placebo

SUMMARY:
In this study, effect of vitamin D supplementation on postoperative pain and sedation-agitation will investigate. Children with mental motor retardation between 7-17 age which dental treatment will be performed under general anaesthesia will be included in this study. 600 IU vitamin D will apply to group D per orally during 12 weeks. Group P will not take anything during 12 weeks. At first day and end of the 12 weeks, serum vitamin D, calcium level will evaluate. At the end of the 12 weeks general anaesthesia will be performed for teeth check up, flouring, scaling polishing, tooth extraction, filling applications, amputations, root canal treatment. After then postoperative pain, sedation and agitation will be evaluate. All data will be statistically evaluate at the end of the study.

DETAILED DESCRIPTION:
Vitamin D deficiency could seem in children with mental and motor retardation. Some researches show that vitamin D supplementations can reduce pain. In this study, the researchers aimed to show effect of vitamin D supplementation on postoperative pain and sedation-agitation. These children which will be applied dental treatment under general anaesthesia included in this study. All subjects randomly divided to the two groups. Every group will include 30 subject. Group D included mentally retarded children which will take daily 600 IU orally vitamin D supplementation during 12 weeks. In the other group(group P) mentally retarded children will not take any supplementation during 12 week. At the first day and last day(after 12 weeks) of study, blood sample will take from all subject. Serum vitamin D, calcium level will evaluate in this sample at the end of the study. All samples will be frozen and stored until testing. All children will be operated under general anaesthesia. Propofol 2mg/kg, rocuronium 0,6 mg/kg will apply for anaesthesia induction. Anaesthesia will maintain with sevoflurane and oxygen- nitrous oxide mixture. Non-communicating Children's Pain Check-list and Ramsey sedation scale will apply all children after postoperative care unit. All children will be evaluate every 15 minutes. After data collection, all data will be analysed with statistically.

ELIGIBILITY:
Inclusion Criteria:

* Mentally and motor retarded children
* dental treatment under general anaesthesia

Exclusion Criteria:

* normally children(not MMR)
* The persons who not accept the including study

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2016-07; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Non-communicating Children's Pain Checklist - Postoperative Version | At Postoperative period for first 1 hour
  The subjects will evaluate per 15 minutes for 1 hour.

SECONDARY OUTCOMES:
vitamin D level | At first day and end of the 12 weeks
  Serum vitamin D level will evaluate At first day and end of the 12 weeks.
Postoperative sedation-agitation | At postoperative first hour
  At postoperative period, every 15 minutes up to 1 hour. Ramsey sedation scores will record.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Ozcengiz, Professor, Study Chair — Cokurova University
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No